CLINICAL TRIAL: NCT05342103
Title: High Flow Nasal Oxygenation Versus Non-invasive Ventilation for Patients With Blunt Chest Trauma: A Comparative Study
Brief Title: High Flow Nasal Oxygenation Versus Non-invasive Ventilation for Patients With Blunt Chest Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huda Fahmy Mahmoud, PhD (Other)
Responsible Party: Sponsor-Investigator, Huda Fahmy Mahmoud, PhD, Assistant professor of Anesthesia and Intensive Care, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 559/9/2021
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-11

CONDITIONS: Chest Trauma
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Intervention Model Description: The patients will be randomly allocated into two groups; patients will receive high-flow nasal oxygenation via nasal cannula (HFNC) or continuous positive airway pressure (CPAP)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal cannula (HFNC) group (Active Comparator): All patients will have FiO2 started at 0.4 and titrated to maintain oxygen saturation (SpO2) ≥ 95%. The flow rate will be set at 60 L/min
  Interventions: Procedure: high flow oxygenation
- Continuous positive airway pressure (CPAP) group (Active Comparator): All patients will have FiO2 started at 0.4 and titrated to maintain oxygen saturation (SpO2) ≥ 95%. Pressure will be set to 3 cm H2O for 5 minutes, then titrated according to patient comfort and tolerance, as well as clinical observation
  Interventions: Procedure: high flow oxygenation

INTERVENTIONS:
Procedure: high flow oxygenation — All patients will have FiO2 started at 0.4 and titrated to maintain oxygen saturation (SpO2) ≥ 95%.

SUMMARY:
Chest trauma remains an issue for health services for both severe and apparently mild trauma management. Severe chest trauma is associated with high mortality and is liable for 25% of mortality in multiple traumas. Moreover, mild trauma is also associated with significant morbidity, especially in patients with preexisting conditions. Thus, whatever the severity, a fast-acting strategy must be organized. In order to improve the prognosis of patients with severe chest trauma, early and continuous application of non-invasive mechanical ventilation (NIV) can indeed reduce the need for intubation and shorten intensive care unit length-of-stay. Among different mechanisms, the early use of positive end-expiratory pressure after chest trauma, when feasible, seems mandatory to optimize oxygenation and improve clinical outcomes. Indeed, interventions aimed at preventing ARDS after chest trauma carry the greatest potential to reduce the substantial morbidity, mortality, and resource utilization associated with this syndrome.

DETAILED DESCRIPTION:
In the past years, High-flow nasal cannula oxygen (HFNC) has gained an important popularity among intensivest to manage patients with acute respiratory failure, filling a gap in the ventilatory support escalation between facemask oxygen and non-invasive or invasive mechanical ventilation. Interestingly, the use of HFNC was widely and rapidly adopted in ICUs.A unique feature of HFNC is its ability to comfortably deliver high flows of warmed humidified gas, 20-70 L min, with a FiO2 range of 0.21-1.0. Physiological responses to HFNC therapy include increases in airway pressure, end-expiratory lung volume (EELV), and oxygenation which are probably optimal with higher flows (60-70 L/min), while the effects on dead-space washout work of breathing, and respiratory rate may be obtained with intermediate flows (20-45 L/min).

Many studies have found that high flow nasal oxygen is much better tolerated by patients compared to non-invasive ventilation, which may improve compliance. Nevertheless, there is no clear consensus on the treatment outcomes (such as intubation rate, escalated respiratory support rate, and mortality) of high flow nasal oxygenation versus non-invasive ventilation for patients with traumatic chest injuries.

ELIGIBILITY:
Inclusion Criteria:

* Rib fractures, pulmonary contusion, and admission within 24 h of injury
* Hypoxemia (SpO2 90 % while breathing 10 l/min oxygen in the ER), or hypercapnia (PaCO2 45 mm Hg) on study entry
* respiratory rate 25/ min despite an optimized intravenous analgesia
* No indication of mechanical ventilation at the time of admission to the intensive care unit

Exclusion Criteria:

* Patients < 18 years old
* Patient already admitted to ICU on mechanical ventilation
* requiring endotracheal intubation and mechanical ventilation immediately on admission for any cause
* facial fractures or base of skull fractures
* Who did not receive a chest computed tomography (CT) scan
* Glasgow Coma Scale ≤ 12

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
the rate of intubation for mechanical ventilation | 48 hours
  Intubation criteria included a respiratory rate of >40 breaths per minute, signs of increased breathing effort, SpO2 of <90% despite high FiO2 or acidosis with a pH of <7.35,occurrence of hemodynamic instability or deterioration of neurologic status.

SECONDARY OUTCOMES:
the Comfort levels with the different modes of oxygen delivery | 48 hours
  will be measured using a 5-point with Likert Scale (marked improvement, slight improvement, no change, slight deterioration, or marked deterioration)
the perceived effort of breathing with the different modes of oxygen delivery | 48 hours
  will be measured using the modified Borg Scale (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Huda Fahmy, Aswān, Egypt